CLINICAL TRIAL: NCT06413550
Title: The Efficacy of Hibiscus Sabdariffa L. Mouth Rinse in Head and Neck Cancer Patients With Xerostomia: A Randomized, Placebo-Controlled Clinical Trial
Brief Title: The Efficacy of Hibiscus Sabdariffa in Xerostomia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Xerostomia & Hibiscus
Record Dates: First submitted 2024-04-19; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Radiation-induced Xerostomia
Keywords: xerostomia; Hibiscus Sabdariffa; Radiation
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): patients in test group will topically apply 20 mL of Hibiscus Sabdariffa L. to the oral mucosa as oral rinse 3 times per day. Patients were advised to rinse 20 mL of Hibiscus Sabdariffa L. from the fourth week of radiotherapy to three months after radiotherapy.
  Interventions: Biological: Hibiscus Sabdariffa
- Control group (Placebo Comparator): Patients in the control arm will topically apply 20 mL of 0.9% of normal saline rinses 3 times per day. Patients were advised to rinse with 20 mL normal saline from the fourth week of radiotherapy to three months after radiotherapy.
  Interventions: Biological: Hibiscus Sabdariffa

INTERVENTIONS:
Biological: Hibiscus Sabdariffa — The fresh red Roselle plant was obtained; the red calyxes of Hibiscus Sabdariffa were separated from the plant and dried for a week at 25°C. The dried calyxes were ground to powder, kept in a sealed container, and stored in a refrigerator (4°C) until used. Aqueous Roselle calyx extract was prepared by adding 10 gm of the previously prepared powder to 100 ml of boiling water and then heated on a hot stirrer plate for 30 min. To remove the remnants, the mixture was filtered via Whatman No 1 filter paper (Whatman products, Springfield Paper Mill, Maidstone, UK). The water content of the filtered solution was evaporated using an air recirculation oven and then kept at 4°C in the dark until used to determine antibacterial effectiveness [20].

SUMMARY:
The goal of this [ type of study: Clinical trial] is to test effectiveness of Hibiscus Sabdariffa L. mouth rinse using the subjective dry mouth score as a primary objective and to assess the effect of that mix on the salivary flow rate and objective dry mouth score as a secondary objective.

DETAILED DESCRIPTION:
Xerostomia, defined as the subjective complaint of dry mouth, is one of the most prevalent and challenging adverse effects for head and neck cancer (HNC) patients treated with radiotherapy (RT) in definitive or adjuvant setting with or without concomitant chemotherapy (CHT). It represents a toxicity that can resolve over time, but often translates into a permanent condition that seriously affects swallowing, speaking and oral health, impairing several domains of patients' quality of life (QoL). Symptomatically, xerostomia may range from mild discomfort to severe oral disease accompanied by signs and symptoms affecting the oral cavity, including mucous membranes, lips, tongue, salivary glands and teeth. In the most severe cases it can cause severe depression.

Although radiation-induced xerostomia (RIX) is multifactorial, it is primarily the consequence of damage to the major and minor salivary glands that are usually included in the radiation fields or are in their close proximity. Thus, the severity of glandular injury and potential for recovery depends on the irradiated gland volume, the cumulative radiation dose and the capability of surviving cells to repopulate. Such injury causes diminution in function of the salivary glands and the consequences are reduction in saliva volume, consistency, pH, immunoglobulins and antimicrobial proteins.

The efficacy of Aqualief in treating xerostomia, or dry mouth, in patients contacting a randomized, placebo-controlled, double-blind trial was evaluated by a previous study. Aqualief contains two key ingredients, carnosine and karkadé (Hibiscus sabdariffa), which were selected and mixed with normalizing saliva pH and increasing saliva buffering activity. These parameters are often impaired in xerostomia patients, leading to acid-induced enamel and dental erosion and promoting the growth of aciduric bacteria.

Aqualief was found to normalize saliva pH to a neutral value and significantly increase the saliva flow rate in xerostomic patients. After six days of treatment, saliva pH was increased toward a neutral value, and the saliva flow rate was increased by almost 60%, compared to the basal value. This improvement was more than three times greater than that achieved with a placebo, which only increased resting salivation by 19%.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, aged above 20 years.
* All patients must have complaint of xerostomia.
* Objective dry mouth score from ( 2-5).
* Subjective dry mouth score from (1-4).
* Patients must be able to make reliable decision or communications.

Exclusion Criteria:

* - Smoking, Alcohol.
* Patient with history of any serious illness as malignancy.
* Patients with any autoimmune disease.
* Vulnerable groups such as pregnant females, prisoners, mentally and physically handicapped individuals.
* Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Subjective symptoms of oral dryness | Three points: -"baseline which is at the fourth week of radiotherapy", -"the second point is at seventh week of the radiotherapy, while the end point is after three months of radiotherapy.
  • Using a questionnaire will be recorded according to the following: Q1. Does your mouth feel dry? Q2. Do you sip liquids to aid in swallowing dry food? Q3. Does your mouth feel dry when eating a meal? Q4. Does the amount of saliva in your mouth seem to be too little? Subject who answered affirmatively to at least one of the questions related to oral dryness will be considered as positive for subjective complaints of oral dryness and take score from 1-4 according to the number of positive answers.
Objective dry mouth score | Three points: -"baseline which is at the fourth week of radiotherapy", -"the second point is at seventh week of the radiotherapy, while the end point is after three months of radiotherapy.
  * The patients will be examined for their signs of dry mouth including:
    1. loss of pooled saliva
    2. Mouth mirror stickiness
    3. Stringy or foamy appearance
    4. Labial dehydration
    5. Irresponsiveness to parotid stimulation
  * Objective dry mouth scores will be calculated as the number of observed dry mouth signs (0-5), and patients with a score less than 2 will be excluded.

SECONDARY OUTCOMES:
Salivary flow rate | Three points: -"baseline which is at the fourth week of radiotherapy", -"the second point is at seventh week of the radiotherapy, while the end point is after three months of radiotherapy.
  • Eating and talking were prohibited during the time of collection. Unstimulated whole saliva will be collected for 5 min by spitting method. The collection will be timed, so that flow rate (mL/min) could be measured.

CONTACTS AND LOCATIONS:
Overall Officials: dalia Ghalwash, Study Director — professor
Locations (1):
- Ahmed Maher Teaching Hosipital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No